CLINICAL TRIAL: NCT01404910
Title: Phase 1b Proof-of-Concept Study of Apheresis to Reduce Soluble Fms-like Tyrosine Kinase-1 (sFlt-1) in Pregnant Women With Preeclampsia Using a Dextran Sulfate Adsorption (DSA) Column (LIPOSORBER® LA-15 System)
Brief Title: Removal of Anti-Angiogenic Proteins in Preeclampsia Before Delivery
Acronym: RAAPID-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Kaneka Medical America LLC (Industry)
Responsible Party: Principal Investigator, Ravi Thadhani, Director of Clinical Research in Nephrology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2012-P-000467/1
Record Dates: First submitted 2011-07-26; First posted 2011-07-28 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Preeclampsia
Keywords: Pregnancy; Preeclampsia; Pre-term; sFlt-1; Apheresis; Hypertension; Proteinuria; VEGF
MeSH Terms: conditions — Pre-Eclampsia; Premature Birth; Hypertension; Proteinuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apheresis (Experimental): Apheresis using Liposorber LA-15 System
  Interventions: Device: Apheresis using Liposorber LA-15 System

INTERVENTIONS:
Device: Apheresis using Liposorber LA-15 System — The Liposorber LA-15 Device is a dextran sulfate cellulose column, one of several currently approved in Europe and United States for pheresis of lipoproteins in the treatment of familial hypercholesterolemia. Such devices have been in use for over 30 years. Published experience in pregnant women with familial hypercholesterolemia suggests that lipoprotein pheresis can be safely used in pregnancy after appropriate individual benefit/risk assessment for both mother and fetus is considered. The Liposorber LA-15 system selected for this trial has been evaluated for its ability to efficiently and selectively remove sFlt-1 in vitro.

SUMMARY:
Preeclampsia is a syndrome that occurs in approximately 3% to 8% of pregnancies and is associated with considerable maternal and neonatal morbidity and mortality. Except for termination of the pregnancy, effective treatments/preventative measures for preeclampsia are lacking. Although prolongation of pregnancy benefits the fetus, it is detrimental to the mother, and is associated with hypertension, proteinuria, and symptoms that suggest kidney, brain, liver and cardiovascular system involvement.

Placental soluble fms-like tyrosine kinase 1 (sFlt-1) is elevated in women with preeclampsia, with levels that fall after delivery. sFlt-1 is a variant of the vascular endothelial growth factor (VEGF) receptor Flt-1, and in the circulation, acts as a potent VEGF and placental growth factor (PlGF) antagonist. Given that sFlt-1 levels are elevated in preeclampsia, we are investigating if removal of sFlt-1 from the plasma of women with preeclampsia can improve maternal and fetal outcomes.

Short-term extracorporeal apheresis with the LIPOSORBER LA-15 System will be the primary intervention using methods that have been previously applied in pregnant women with familial hypercholesterolemia.

DETAILED DESCRIPTION:
The primary objective of this trial is to determine whether short-term apheresis using a dextran sulfate adsorption (DSA) column (Liposorber LA-15 System; the Device) leads to a reduction in circulating sFLT-1 in the blood of women with pre-term preeclampsia.

The following secondary objectives are aimed at evaluating the efficacy and safety of the Device as well as the impact of removing circulating sFlt-1 on maternal and neonatal outcomes:

1. To determine whether short-term apheresis using the Device in women with pre-term preeclampsia leads to:

   * a prolongation of pregnancy (ie, gestational age)
   * a reduction in blood pressure (BP) and proteinuria
   * an increase in fetal birth weight
2. To determine the safety of reducing maternal sFlt-1 levels using the Device.

Up to 16 patients will be enrolled. Initially, 4 patients will undergo apheresis UP TO 2 times in the first week and undergo all protocol-related assessments including PK of sFlt-1 levels. Based on an assessment of clinical response by the Investigator, these first 4 patients will be offered the option to continue apheresis treatments (without pharmacokinetic [PK] assessments) up to twice weekly until delivery or until 34 weeks gestation, whichever comes first. Following complete review of all parameters and outcomes by an independent Data Safety Monitoring Board (DSMB), up to 12 additional patients will be enrolled (total of up to 16).

UPDATE: The DSMB reviewed data after the first 4 patients and again after 10 patients/delivered infants had been treated. In the next 6 patients, DSMB review will occur after every 3 patients/delivered infants. These remaining 6 patients may undergo apheresis up to 3 times per week.

ELIGIBILITY:
Inclusion Criteria (maternal):

1. Signed informed consent in a pregnant woman ages 18 and 45 years hospitalized for pre-term preeclampsia
2. Pre-term preeclampsia defined by systolic BP ≥140 mm Hg or ≥90 mm Hg diastolic at or after 23 weeks of gestation or at or before 32 weeks in gestation in a woman with previously normal BP and proteinuria 0.3 grams in a 24-hour specimen or urine protein/creatinine ratio >0.30.
3. sFlt-1/PlGF ratio >85 (blood levels of sFlt-1 and PlGF determined using CE-approved Roche Diagnostics assays).

Exclusion Criteria (Maternal and Fetal):

Maternal:

1. Taking any form of angiotensin cascade blocker
2. History or diagnosis of pre-existing chronic hypertension (first 3 patients only)
3. History of cardiac impairments including uncontrolled arrhythmia, unstable angina, decompensated congestive heart failure or valvular disease
4. History or diagnosis of chronic renal disease
5. Patients receiving anticoagulation therapy prior to study entry
6. Anticipated immediate delivery within 24 hours
7. Signs of central nervous system (CNS) dysfunction, including seizures, cerebral edema (CT-scan or MRI)
8. History of thyroid disease
9. History of liver abnormalities
10. Pulmonary edema
11. Thrombocytopenia (platelet count < 100,000/mm3)
12. Anemia - hemoglobin < 8 g/dL
13. Evidence of "reverse Doppler" flow on umbilical Doppler
14. Placenta previa
15. Placental abruption
16. Pre-term labor
17. Active hepatitis B, C, or tuberculosis infection or HIV positive status
18. Any condition that the investigator deems a risk to the patient or fetus in completing the study.
19. Any condition which in the opinion of the investigator would necessitate delivery in the next 24 hours

Fetal characteristic that would exclude the mother from participating:

1. Trisomy
2. Biophysical profile (BPP) < 6
3. Amniotic fluid index (AFI) < 5 cm
4. Estimated fetal weight (EFW) < 5th percentile for gestational age (IUGR)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2013-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
sFlt-1 levels measured immediately prior to each apheresis treatment, and at 2-4, 12, 24, etc. (every 24 hours) following termination of apheresis to determine kinetics of sFlt-1 clearance (until delivery). | 12 months
  The study period for each patient will be from initiation of the device until 30 days (± 7 days) after delivery. Additional assessments will be performed at 90 and 365 days (± 7 days, respectively) using maternal and neonatal medical records and/or by telephone contact with the mother.

SECONDARY OUTCOMES:
Maternal and fetal safety | 12 months
  Maternal: Blood pressure, proteinuria, coagulation parameters, elevated liver enzymes, and low platelet count (HELLP) syndrome, maternal complications Fetal: Early fetal assessments delivery (birth) will include gestational age, birth weight, length, fetal APGAR scores (1'/5'/10'), amniotic fluid volume by ultrasonography, and head circumference, NICU details, pulmonary parameters and any neonatal complications (eg, ventilatory support, respiratory distress syndrome, CRIB-Score, cerebral hemorrhage, ischemic colitis, and retinopathy of prematurity [ROP]) and compared to historical milestones. Fetal cord blood (with maternal consent) is to be sampled from umbilical artery at delivery to determine sFlt-1 levels, to measure pH and stored for later biochemical analyses. Fetal assessments will also occur ~30, 60, 90 and 365 days after delivery.
Maternal and fetal efficacy | 12 months
  Maternal:
  Prolongation of pregnancy, reduction in blood pressure and proteinuria
  Fetal:
  Outcomes will be collected on all births, at birth, 24-hours post-partum, 72-hours post-partum, 30 day status vs historical milestones. 90 and 365 day assessments will be made using data obtained from medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi I Thadhani, MD, MPH, Principal Investigator — Massachusetts General Hospital; Thomas Benzing, MD, Principal Investigator — University of Koln; Holger Stepan, MD, Principal Investigator — University of Leipzig
Locations (3):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- Germany (2):
  - University Hospital of Cologne (Universitat zu Koln), Cologne
  - University Hospital Leipzig, Leipzig

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thadhani R, Kisner T, Hagmann H, Bossung V, Noack S, Schaarschmidt W, Jank A, Kribs A, Cornely OA, Kreyssig C, Hemphill L, Rigby AC, Khedkar S, Lindner TH, Mallmann P, Stepan H, Karumanchi SA, Benzing T. Pilot study of extracorporeal removal of soluble fms-like tyrosine kinase 1 in preeclampsia. Circulation. 2011 Aug 23;124(8):940-50. doi: 10.1161/CIRCULATIONAHA.111.034793. Epub 2011 Aug 1. PMID 21810665
- [Background] Easterling TR. Apheresis to Treat Preeclampsia: Insights, Opportunities and Challenges. J Am Soc Nephrol. 2016 Mar;27(3):663-5. doi: 10.1681/ASN.2015070794. Epub 2015 Sep 24. No abstract available. PMID 26405110
- [Result] Thadhani R, Hagmann H, Schaarschmidt W, Roth B, Cingoez T, Karumanchi SA, Wenger J, Lucchesi KJ, Tamez H, Lindner T, Fridman A, Thome U, Kribs A, Danner M, Hamacher S, Mallmann P, Stepan H, Benzing T. Removal of Soluble Fms-Like Tyrosine Kinase-1 by Dextran Sulfate Apheresis in Preeclampsia. J Am Soc Nephrol. 2016 Mar;27(3):903-13. doi: 10.1681/ASN.2015020157. Epub 2015 Sep 24. PMID 26405111